CLINICAL TRIAL: NCT02989441
Title: Peripheral Perfusion Index as Marker for Systemic Hemodynamics During Anesthesia
Brief Title: Perfusion Index in Anesthesia
Status: Completed | Type: Observational
Sponsor: Jakob Højlund (Other)
Responsible Party: Sponsor-Investigator, Jakob Højlund, Medical Doctor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: H-16030081
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Monitoring, Physiological
Keywords: Perfusion Index; Hemodynamics; Anesthesia; Stroke Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In patients under general anesthesia the investigators wish to investigate association and covariance between a peripheral perfusion index as obtained by Radical 7 monitor (Masimo, Irvine, CA, USA) and more traditional hemodynamic parameters, ie. invasive blood pressure and SV as obtained by LiDCO rapid monitor (LiDCO Ldt., London, UK)

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective and sub-acute surgical repair of para-oesophagal hernia.
* Willingness to participate

Exclusion Criteria:

* Patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for elective and sub-acute surgical repair of para-oesophagal hernia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Co-variance between Perfusion Index (PI) and Cardiac Output (CO) and Stroke Volume (SV) | Intra-operative

SECONDARY OUTCOMES:
Co-variance between Perfusion Index (PI) and Mean Arterial Pressure (MAP) | Intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD PhD, Study Chair — Hvidovre University Hospital, University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided